CLINICAL TRIAL: NCT07131371
Title: Stratification, Management, and Guidance of Hypertrophic Cardiomyopathy Patients Using Hybrid Digital Twin Solutions
Acronym: SMASH-HCM
Status: Active, not recruiting | Type: Observational
Sponsor: Tampere University (Other)
Collaborators: University of Bologna (Other); Universita Degli Studi di Firenze (Unknown); Rennes University Hospital (Other); University of Milan (Other); University College Dublin (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Medtronic Bakken Research (Industry); Pharmatics Limited (Unknown); University of Oxford (Other); University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Katriina Aalto-Setälä, Professor, Tampere University
Other Study IDs: 101137115
Record Dates: First submitted 2025-07-10; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: HCM - Hypertrophic Cardiomyopathy
Keywords: HCM; digital twin; AI; in silico modelling; iPSC-derived cardiomyocytes
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCM patients from Florence Italy, Rennes, France, and Tampere Finland: HCM patients in follow up

SUMMARY:
The goal of SMASH-HCM is to develop a digital twin or virtual model of the heart and vascular system with sympathetic nerve control that integrates multi-scale and multi-organ spatiotemporal biophysical data from a multitude of sources. SMASH-HCM's digital twin powered platform will dramatically improve hypertrophic cardiomyopathy (HCM) patient stratification and disease management through stepwise deep phenotyping integrated in clinical and patient-guided workflows.

DETAILED DESCRIPTION:
The aim of this SMASH-HCM study is with available well-characterized clinical data and existing iPSC derived cardiomyocyte data from HCM patients to find better predictors of worse outcomes i.e. potentially lethal arrhythmias, heart failure, sudden cardiac arrest in HCM patients. Additionally with artificial intelligence (AI) to find markers of good outcome so that we could focus more on those who would potentially benefit more from the intense follow up. Additionally our aim is to create a digital twin by collecting all possible clinical data from the HCM patients and also from currently healthy mutation carriers to be able to predicts the clinical out in more personal way and also toddling treatment strategies in more personal manner.

ELIGIBILITY:
Inclusion Criteria:

* HCM or carrying. mutation for HCM

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCM patients followed in the clinical sites in this study: Florence Italy, Rennes France and Tampere Finland
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of patients with severe arrhythmias, heart failure, sudden death or implantation of ICD for Digital Twin creation | from patient records until the end of 2026
  The presence of arrhythmias will be obtained from 24 h Holter recordings, stress exercise test, monitor recording if in the hospital and if found in clinical patient records.
  Heart failure data if obtained from ultrasound records, clinical observations and elevated natriuretic peptide levels in the serum.
  Data about sudden deaths are obtained from patient records. Requirements of ICD implantations are obtained from patient records

OTHER OUTCOMES:
Other clinical characteristics of patients with severe outcomes due to HCM compared to those with mild disease for the creation of SMASH-HCM algorithm. | January 2024 to December 2026
  All cardiac medication will be recorded and the reason this has changed during the analysis timepoints.
  Incidence of other diseases will be included in the analysis e.g. stroke, myocardial infarction, atrial fibrillation, depression, changes in vascular status (mainly blood pressure) The number of hospital visits is recorded and the reason for those

CONTACTS AND LOCATIONS:
Overall Officials: Jari Hyttinen, Professor, Study Director — Professor
Locations (1):
- Tampere university, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
Clinical data (ECG, ultra sound, cardiac MR, cardiac biomarkers, gene mutations, additional diseases) found in patient files will be shared with this study consortium with different AI groups specializing in each specific clinical record.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1.1.2025-31.12.2028
Access Criteria: The databank is simply a file-sharing app using Nextcloud, with user access controls and monitoring
URL: https://smash-hcm.ucd.ie/login